CLINICAL TRIAL: NCT03665428
Title: Helicobacter Pylori Eradication Rates of Bismuth-containing Quadruple Therapy vs Modified Quadruple Therapy in Korea; Open-label, Randomized Controlled Trial
Brief Title: Helicobacter Pylori Eradication Rates of Bismuth-containing Quadruple Therapy vs Modified Quadruple Therapy in Korea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Collaborators: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Chang Seok Bang, Associate professor of Hallym University College of Medicine, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSBang2018HP
Record Dates: First submitted 2018-06-25; First posted 2018-09-11 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: helicobacter pylori infection; Drug Resistance, Microbial

STUDY DESIGN:
Intervention Model Description: PAMB group (modified quadruple therapy) vs. PBMT group (bismuth-containing quadruple therapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAMB group (Experimental): PAMB treatment (modified quadruple therapy) for 14 days
  Interventions: Drug: PAMB treatment (modified quadruple therapy)
- PMBT group (Active Comparator): PBMT treatment (bismuth-containing quadruple therapy) for 14 days
  Interventions: Drug: PBMT treatment (bismuth-containing quadruple therapy)

INTERVENTIONS:
Drug: PAMB treatment (modified quadruple therapy) — Randomly assign either as PAMB or PBMT group treatment
  Other Names: PBMT treatment (bismuth-containing quadruple therapy)
  Arms: PAMB group
Drug: PBMT treatment (bismuth-containing quadruple therapy) — Randomly assign either as PAMB or PBMT group treatment
  Other Names: PAMB treatment (modified quadruple therapy)
  Arms: PMBT group

SUMMARY:
South Korea has the highest incidence of gastric cancer worldwide and Helicobacter pylori infection is still prevalent. Clarithromycin-containing triple therapy is still the primary therapy approved by the Korean government. However, studies of antibiotic resistance has shown that regional resistance pattern to antibiotics such as clarithromycin, metronidazole, or quinolone. Recent study in Korea has shown that modified-quadruple therapy has comparable eradication rate to concomitant therapy. However, there has been no comparable study of modified-quadruple therapy with bismuth-containing quadruple therapy. The aim of this study is to compare the eradication rate of modified-quadruple therapy and bismuth-containing quadruple therapy with presenting phenotypic and genotypic antibiotic resistance profile.

DETAILED DESCRIPTION:
South Korea has the highest incidence of gastric cancer worldwide and Helicobacter pylori infection is still prevalent. Clarithromycin-containing triple therapy is still the primary therapy approved by the Korean government. However, studies of antibiotic resistance has shown that regional resistance pattern to antibiotics such as clarithromycin, metronidazole, or quinolone. Recent study in Korea has shown that modified-quadruple therapy has comparable eradication rate to concomitant therapy. However, this study did not explore the antibiotic resistance profile of Helicobacter pylori. And, there has been no comparable study of modified-quadruple therapy with bismuth-containing quadruple therapy. The aim of this study is to compare the eradication rate of modified-quadruple therapy and bismuth-containing quadruple therapy with presenting phenotypic and genotypic antibiotic resistance profile.

ELIGIBILITY:
Inclusion Criteria:

* Participants who had upper endoscopic examination within 3 months and diagnosed by Helicobacter pylori infection either by rapid urease test, urea breath test, or histopathologic examination.
* Participants who voluntarily want to participate in this study.

Exclusion Criteria:

* Participants who had history of Helicobacter pylori eradication.
* Participants who had experience of stomach resection.
* Participants who had history of allergy or adverse events related to eradication medication.
* Participants who had history of administration of proton-pump inhibitor within 2 weeks or Histamine 2 receptor blocker within 1 week.
* Participants who had history of administration of these drugs within a week or who need continuous administration of these drugs; aspirin (except low-dose aspirin for primary prophylaxis of cardiovascular disease), intravenous or oral NSAID, anticholinergics, prostaglandin analogs, pro-motility drugs, sucralfate
* Participants who had history of administration of antibiotics within 4 weeks.
* Pregnant, breast feeding participant or who do not have a will to avoid pregnancy during clinical trial
* Participants who are administrating one of these drugs (Lovastatin, Simvastatin, Atorvastatin, Indinavir, Ritonavir, Cyclosporin, Terfenadine, Cisapride, Pimozide, Astemizole, HIV protease inhibitors (Atazanavir, Nelfinavir), Ergotamine, Dihydroergotamine, Mizolastine, Bepridil, Ticagrelor)
* Participants who have infectious mononucleosis, central nervous system infection, hematologic disease, galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption, Torsades de pointes.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of eradication success | up to 4 weeks
  Eradication success means negative urea breath test done at least after 4 weeks from medication administration

SECONDARY OUTCOMES:
Rate of adverse events related to eradication medication | up to 4 weeks
  Adverse events related to eradication medication
Rate of compliance of eradication medication administration | up to 4 weeks
  Compliance (percentage of amount) of eradication medication administration

CONTACTS AND LOCATIONS:
Overall Officials: Chang Seok Bang, MD, PhD, Principal Investigator — Hallym University
Locations (1):
- Chuncheon Sacred Heart hospital, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No